CLINICAL TRIAL: NCT02773602
Title: Effect of Dexamethasone or Clonidine When Given as Adjuncts to Ropivacaine for Caudal Analgesia on Duration of Analgesia Compared to Placebo in Children
Brief Title: Dexamethasone or Clonidine as Adjuncts to Ropivacaine for Caudal Analgesia on Analgesia Duration in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor of pediatric Anesthesia, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-11-0002
Record Dates: First submitted 2015-12-11; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
Keywords: Analgesia; caudal analgesia; ropivacaine; clonidine; dexamethasone
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexamethasone; Clonidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexamethasone (Experimental): Dexamethasone has been used for adult epidurals and nerve blocks and in spine surgeries. It prolongs the duration of pain relief and causes less sedation. It is commonly administered to children during surgery to help decrease nausea and vomiting after surgery. It is also much cheaper than clonidine The patient will receive Ropivacaine plus 200 μgm/kg of dexamethasone in 1 ml saline
  Interventions: Drug: Dexamethasone
- Clonidine (Active Comparator): Clonidine has been added to caudal analgesia for infants and children for many years. It increases the duration of pain relief of ropivicaine by itself, however, it may lead to prolonged sedation following the surgical procedure (an undesired effect) and it is expensive.
  The patient will receive Ropivacaine plus 2 μg/kg of clonidine in 1 ml saline.
  Interventions: Drug: Clonidine
- Normal Saline (Placebo Comparator): The patient only will receive Ropivacaine
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — 200 μgm/kg of dexamethasone in 1 ml saline
  Arms: Dexamethasone
Drug: Clonidine — 2 μg/kg of clonidine in 1 ml saline
  Arms: Clonidine
Drug: Normal Saline — 1 ml of saline added to the ropivacaine, 0.2%, 1 ml/kg
  Arms: Normal Saline

SUMMARY:
Comparing the duration of pain relief from caudal analgesia when adjuncts like dexamethasone, clonidine, or saline (salt water) are added to ropivacaine.

DETAILED DESCRIPTION:
The local anesthetic, which is currently used for caudal analgesia, is called ropivacaine. It works well and is safe in infants and children. Doctors commonly add small amounts of other medication to ropivacaine to prolong the duration of pain relief provided by a single injection of caudal analgesia.

In this study, the length of duration of pain relief the child receives from caudal analgesia will be examined when different medications are added to ropivacaine. Specifically, dexamethasone, clonidine, or saline (salt water) will be added to ropivicaine and the length of time it takes before the child needs more pain medication will be determined.

Clonidine has been added to caudal analgesia for infants and children for many years. It increases the duration of pain relieving effect of ropivicaine by itself, however, it may lead to prolonged sedation following the surgical procedure (an undesired effect) and it is expensive.

Dexamethasone has been used for adult epidurals and nerve blocks and in spine surgeries. It prolongs the duration of pain relief and causes less sedation. It is commonly administered to children during surgery to help decrease nausea and vomiting after surgery. It is also much cheaper than clonidine.

ELIGIBILITY:
Inclusion Criteria:

* The subject will receive presurgical caudal block
* American Society of Anesthesiologists (ASA) 1 or 2
* Day surgery unit
* weight 30 kg or less

Exclusion Criteria:

* Neuromuscular disease
* Back problem
* Caudal area skin infection
* Mental retardation
* Developmental delay
* Bleeding disorder

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Duration of block | Within 24 hours after surgery
  Duration of block is calculated from time of first pain medication minus time of caudal placement. Caudal placement occurs before pain medication is administered.

SECONDARY OUTCOMES:
Number of children between the groups who received pain medication in the PACU | Within 24 hours after surgery
Number of children between the groups who received pain medication after hospital discharge | Within 24 hours after surgery
number of children group between the groups who required pain medication in first 24 h after surgery | Within 24 hours after surgery
Awakening time | Within 24 hours after surgery
  Awakening time is calculated from the end of anesthesia to time to reach Steward Score of 6. Patients who are awake, coughing/crying, and have purposeful movements are assigned a Steward Score of 6.

CONTACTS AND LOCATIONS:
Overall Officials: Samia N Khalil, (M.B; B.CH), Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States